CLINICAL TRIAL: NCT00001908
Title: T Cell Cytokine Changes During IL-4 Receptor Treatment for Asthma
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990114; 99-I-0114
Record Dates: First submitted 1999-11-03; First posted 2002-05-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-07

CONDITIONS: Asthma; Hypersensitivity
Keywords: Allergy; Interleukin; Immunomodulator; Th2; Inflammation; Asthma
MeSH Terms: conditions — Asthma; Hypersensitivity; Inflammation

SUMMARY:
Asthma is a chronic inflammatory disorder of the airways characterized by reversible airflow obstruction. Fourteen million people (6.4%) in the United States report having asthma, and from 1980 to 1994 the prevalence of self-reported asthma in the United States increased 75%. Interleukin-4 (IL-4) plays a key role in this response by promoting IgE production, upregulating IgE receptors, upregulating adhesion receptors such as VCAM-1, promoting Th2 cell development and promoting mucus secretion. A soluble form of the receptor for IL-4 (IL-4R) that has antagonist activity has been developed for clinical use. Soluble IL-4R acts by competing with endogenous cell bound IL-4R for free IL-4, thus inhibiting IL-4 function. IL-4 is required for the development of allergen specific Th2 memory cells. Less well understood are the factors required for maintenance of Th2 responses. The maintenance of polarized Th2 responses to allergens have been postulated to require IL-4 itself, by acting as an anti-apoptotic/survival factor or by differentiating naive allergen specific T cells to the Th2 phenotype. Subjects on sIL-4 therapy represent a unique patient group that possess allergen specific Th2 cells, but in which the capacity for IL-4 to promote further Th2 cell survival or differentiation has been blocked. This is a single site adjunct study proposed to study subjects ages 14 years and older who are enrolled at the NIH Clinical Center on a multicenter trial of IL-4R in moderate to severe asthma (Phase II Efficacy Study of Aerosolized Recombinant Human IL-4 Receptor in Asthma). A maximum of 40 subjects will be enrolled. We hypothesize that effective blocking of such Th2 priming would result in a decreased frequency of both allergen specific Th2 cells as well as mitogen activated Th2 cells. Determination of the fate of Th2 cell responses during long term IL-4R therapy may have important implications both for future development of anti-cytokine therapies as well as for understanding the T cell biology of allergic diseases and asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways characterized by reversible airflow obstruction. Fourteen million people (6.4%) in the United States report having asthma, and from 1980 to 1994 the prevalence of self-reported asthma in the United States increased 75%. Interleukin-4 (IL-4) plays a key role in this response by promoting IgE production, upregulating IgE receptors, upregulating adhesion receptors such as VCAM-1, promoting Th2 cell development and promoting mucus secretion. A soluble form of the receptor for IL-4 (IL-4R) that has antagonist activity has been developed for clinical use. Soluble IL-4R acts by competing with endogenous cell bound IL-4R for free IL-4, thus inhibiting IL-4 function. IL-4 is required for the development of allergen specific Th2 memory cells. Less well understood are the factors required for maintenance of Th2 responses. The maintenance of polarized Th2 responses to allergens have been postulated to require IL-4 itself, by acting as an anti-apoptotic/survival factor or by differentiating naive allergen specific T cells to the Th2 phenotype. Subjects on sIL-4 therapy represent a unique patient group that possess allergen specific Th2 cells, but in which the capacity for IL-4 to promote further Th2 cell survival or differentiation has been blocked. This is a single site adjunct study proposed to study subjects ages 14 years and older who are enrolled at the NIH Clinical Center on a multicenter trial of IL-4R in moderate to severe asthma (Phase II Efficacy Study of Aerosolized Recombinant Human IL-4 Receptor in Asthma). A maximum of 40 subjects will be enrolled. We hypothesize that effective blocking of such Th2 priming would result in a decreased frequency of both allergen specific Th2 cells as well as mitogen activated Th2 cells. Determination of the fate of Th2 cell responses during long term IL-4R therapy may have important implications both for future development of anti-cytokine therapies as well as for understanding the T cell biology of allergic diseases and asthma.

ELIGIBILITY:
Patients must be 14 years of age or older.

Must be participating in 99-I-0115 "Phase II Efficacy Study of Aerosolized Recombinant Human IL-4 Receptor in Asthma".

If younger than 18 years old, must weigh 50 kg or more.

Must have HIV seronegativity.

Must not have hemoglobin less than 12 g/dL.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1999-06; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Savelkoul HF, van Ommen R. Role of IL-4 in persistent IgE formation. Eur Respir J Suppl. 1996 Aug;22:67s-71s. PMID 8871047
- [Background] Paul WE, Seder RA. Lymphocyte responses and cytokines. Cell. 1994 Jan 28;76(2):241-51. doi: 10.1016/0092-8674(94)90332-8. No abstract available. PMID 7904900
- [Background] Boise LH, Minn AJ, June CH, Lindsten T, Thompson CB. Growth factors can enhance lymphocyte survival without committing the cell to undergo cell division. Proc Natl Acad Sci U S A. 1995 Jun 6;92(12):5491-5. doi: 10.1073/pnas.92.12.5491. PMID 7777536